CLINICAL TRIAL: NCT04154241
Title: Developing a Method Using PET-MR to Improve Staging and Monitoring of Neuroendocrine Tumor
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TASMC-19-ES-0583-CTIL
Record Dates: First submitted 2019-10-29; First posted 2019-11-06 (Actual); Last update posted 2019-11-06 (Actual); Status verified 2019-11

CONDITIONS: Neuroendocrine Tumors
MeSH Terms: conditions — Neuroendocrine Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- neuroendocrine tumor Patients (Experimental): A cohort of patients that were diagnosed with NET using biopsy.
  Interventions: Diagnostic Test: PET/MR scan

INTERVENTIONS:
Diagnostic Test: PET/MR scan — The PET will be performed with (68Ga)-labeled somatostatin analogue since it was proven to be superior to other NET PET tracers in terms of lesion detection and sensitivity [11] [12]. The 3 tesla magnet of the MRI should allow acquisition of several contrasts within a reasonable time frame. The protocol will include T1 and T2-weighted images, diffusion-weighted images with multiple b values and apparent diffusion coefficient (ADC) maps.
  All images will be analyzed with big data tools such as radiomics and texture analysis in order to integrate all image parameters and different contrasts into individual tumor status. Then, accuracy, sensitivity and specificity will be evaluated by correlation of this data collection and analysis method with histological biomarkers (for example, Ki67 level) and treatment results.

SUMMARY:
euroendocrine tumors (NETs) are neoplasms that originate from diffuse neuroendocrine system which consist about 17 types of different neuroendocrine cells. These cells combine properties of nerve cells with properties of endocrine cells, that is they receive neuronal signal and produce hormones.The most common locations for NETs are the lungs and organs of the gastroenteropancreatic (GEP) system, however they can be found in any other organ in the body . Clinically, functional NET cells secrete hormones which cause symptoms such as diarrhea or flushing, however non-functional NET cells also exist posing a challenge in the identification and diagnosis of the disease . Besides surgery to remove the tumor, there are numerous of treatment options for systemic handling of the NETs. These treatments include: somatostatin analogues, interferon, chemotherapy, transarterial (chemo) embolisation, radiofrequency ablation, sunitinib, everolimus and radionuclide targeted therapy. The choice of treatment depends on the correct characterization of the NET, primary tumor location, tumor subtype, grade and stage of the disease . Biomarkers for NETs serve a critical role in the diagnosis stage, where it is highly important to identify the NET type and precise location. Furthermore, selecting the correct biomarkers for monitoring the disease is important to predict response for treatment and allow the choice of the right treatment from the large variety of treatment options. NET biomarkers include circulating biomarkers such as Chromogranin A, Ki67, Neuron Specific Enolase (NSE), 5 hydroxyindoleacetic acid (5HIAA) and many others found in blood samples, or in the tumor tissue . Beside the circulating biomarkers, imaging biomarkers plays a central role in diagnosis, staging, treatment selection and follow-up of NETs . Current imaging tools are morphological modalities such as CT, MRI and Ultrasound and molecular imaging. Several types of molecular imaging techniques are performed to characterize NETs: single photon emission computed tomography (SPECT) with 111In-pentetreotide, largely superseded now by positron emission tomography (PET) with 68Ga-labeled somatostatin analogs, is used to identify the somatostatin receptor status.

DETAILED DESCRIPTION:
18F-DOPA and 11C-5-HTP are used to evaluate neuroendocrine metabolism . 18-fluoro-deoxy-glucose (FDG) PET is usually a poor indication for NETs since these neoplasms tend to be metabolic inactive, and thus FDG-PET is only used for high grade more aggressive NETs . Only a combination of several biomarkers together can lead to NET description that allows treatment selection and to some extent prediction of treatment success.

In this study the investigators wish to take advantage of the new hybrid PET-MR and use it to find new methods to characterize NETs. Only very few PET-MR studies have been performed with correlation to NETs and they showed the potential of this tool for tumor characterization .

The investigators plan to integrate PET-MR with big data analysis methods to obtain an improved tool for staging, characterization and monitoring NETs.

ELIGIBILITY:
Inclusion Criteria:

A cohort of patients that were diagnosed with NET using biopsy.

Exclusion Criteria:

1. Age <18.
2. Pregnant or breast feeding patients.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-03-10 (Estimated); Primary Completion 2021-05-10 (Estimated); Study Completion 2022-03-10 (Estimated)

PRIMARY OUTCOMES:
Patients who preformed PET/MR. | 1 year
  The investigators develop new methods for the characterization and monitoring of NETs using the latest state of the art PET-MR technology combined with big data analysis methods in order to obtain a more accurate, specific and sensitive biomarker.

IPD SHARING:
Plan to Share IPD: Undecided